CLINICAL TRIAL: NCT00892515
Title: Women In Steady Exercise Research (WISER) Sister
Brief Title: Exercise Programs in Healthy Young Women at Increased Risk of Developing Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: CDR0000617105; UPCC-807822; UPCC-09108
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Healthy, no Evidence of Disease
Keywords: breast cancer; healthy, no evidence of disease
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling; Chromatography, Gas; Immunoenzyme Techniques; Immunologic Techniques; Mass Spectrometry; Absorptiometry, Photon; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental)
  Interventions: Behavioral: exercise intervention; Other: counseling intervention; Other: gas chromatography; Other: immunoenzyme technique; Other: immunologic technique; Other: laboratory biomarker analysis; Other: mass spectrometry; Other: physiologic testing; Other: questionnaire administration; Other: survey administration; Procedure: dual x-ray absorptometry; Procedure: magnetic resonance imaging; Procedure: study of high risk factors

INTERVENTIONS:
Behavioral: exercise intervention
Other: counseling intervention
Other: gas chromatography
Other: immunoenzyme technique
Other: immunologic technique
Other: laboratory biomarker analysis
Other: mass spectrometry
Other: physiologic testing
Other: questionnaire administration
Other: survey administration
Procedure: dual x-ray absorptometry
Procedure: magnetic resonance imaging
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Exercise may change the risk of developing breast cancer. It is not yet known whether low-intensity exercise or high-intensity exercise is more effective in lowering the risk of breast cancer.

PURPOSE: This randomized clinical trial is studying how well exercise programs work in healthy young women at increased risk of developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To conduct a dose response study of low- or high-dose exercise over 5 menstrual cycles, with no concomitant dietary changes producing a caloric deficit, in healthy younger women with ≥ 18% lifetime risk for developing breast cancer.
* To determine the effects of this exercise regimen on variables known to be associated with breast mitotic activity in these participants.

Secondary

* To assess changes in other physiologic parameters associated with breast mitotic activity (i.e., urinary progesterone [pregnanediol-glucuronide, PdG] from daily first morning urine samples; follicular phase circulating [serum] levels of estradiol, progesterone, testosterone, and prolactin; follicular phase breast density [fibroglandular tissue volume] from magnetic resonance imaging; estrogen metabolites [estrone, estradiol, estriol, 2-OHE_1, 2-OHE_2, 4-OHE_1, 4-OHE_2, 16-OHE_1 and ratios]; adipokines [i.e., adiponectin and Leptin]; and body composition [i.e., % body fat, lean mass, fat mass, total mass]) in these participants.
* To assess the extent to which changes in body composition and/or body mass mediate observed changes in these participants.
* To quantify the relationship between estrogen and progesterone from daily urinary measurements with observed menstrual cycle alterations such as follicular and luteal phase length changes, and ovulatory status in these participants.
* To compare levels and exercise-induced changes in urinary estrogens, estrogen metabolites, circulating hormones, adipokines, and body size across two groups of women who differ as to breast cancer risk in an exploratory manner.

OUTLINE: Patients are stratified according to body mass index (21-29.9 vs 30-50) and gynecologic age (< 10 vs ≥ 10 years since start of menstruation). Participants are randomized to 1 of 3 intervention arms.

* Arm I (control): Participants are placed on a waiting list to receive the exercise intervention at completion of the study.
* Arm II: Participants undergo a low-intensity exercise program comprising 150 minutes of exercise per week for 20 weeks. They are given a treadmill at the beginning of the study and offered ongoing support from a certified exercise professional. Participants may exercise at home on the provided treadmill or at a gym of their choosing. Participants must maintain weekly contact with the exercise professional for the duration of the study, either by phone for brief phone counseling or at a weekly group exercise session at a participating YMCA. The exercise professional visits the participant's home for the first exercise session of each of the first 5 weeks to help individualize the intensity and duration of the exercise session and to instruct participants on the use of the exercise logs and on injury prevention.

Exercise intensity is measured by a Polar Heart Rate monitor worn by the participant to record heart rate response during exercise. Every two weeks, the exercise professional reviews downloadable heart-rate data from the monitor during the home or group exercise session, to objectively measure exercise adherence and provide guidance and emotional support to the participant.

* Arm III: Participants undergo a high-intensity exercise program that begins with 150 minutes of exercise per week and then gradually builds to 300 minutes per week over 10 weeks. Participants continue to exercise at the higher level until the end of the 20-week intervention period. Participants also undergo exercise and heart rate monitoring and brief phone counseling as in arm II.

Blood and urine samples are obtained from participants periodically before and/or during study to evaluate factors associated with breast mitotic activity and linked to breast cancer risk: urinary conjugates (i.e., E1G and PdG) by enzyme immunoassays; urinary estrogen metabolites by gas chromatography/mass spectrometry; circulating hormones (i.e., estradiol, progesterone, testosterone, and prolactin) by radioimmunoassay; and adipokines (i.e., adiponectin and leptin) by sandwich ELISA. Participants also undergo physical assessments, including periodic measures of body composition by DEXA, follicular phase breast density (fibroglandular tissue volume) by MRI, and height and weight. Aerobic fitness and physical activity levels are also assessed.

Participants complete surveys and questionnaires periodically during study to obtain information on demographics, health history, medication use, eating disorders, dietary intake, and menstrual history.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy women with ≥ 18% lifetime risk for breast cancer as evidenced by the following:

  * Documentation from a genetic counselor of a known familial breast cancer susceptibility mutation
  * Claus model risk of ≥18%
  * Predicted probability of BRCA1/2 mutation > 25% based on the Myriad model
  * Documentation of a known mutation in a family member such that the Mendelian probability of a BRCA1/2 mutation would be >25%
  * History of lobular carcinoma in situ
* No prior prophylactic mastectomy
* Leisure-time exercise energy expenditure of ≤ 500 kcal/week over the past 6 months
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Premenopausal
* Menstrual cycles 25-32 days in length
* Intact ovaries and uterus
* Gynecologic age (defined as participant's current age minus the age at which she started menstruating) of at least 4 years
* Body mass index 21-50
* No history of menstrual difficulties
* No history of physician-diagnosed gynecological disease (e.g., fibroids, endometriosis, or polycystic ovary syndrome)
* Not pregnant
* Not planning to become pregnant during the study period
* No medical conditions or medications that would prohibit participation in aerobic exercise or would negatively impact the study
* No history of cancer, except nonmelanoma skin cancers, and in situ cervical cancers
* No eating disorders (e.g., bulimia or binge-eating disorder)
* At least one year since prior smoking
* Not planning to move away from the area during the period of the study
* No concurrent participation in any weight loss programs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 months since prior hormonal contraception
* Must use effective non-hormonal contraception unless participant has undergone prior tubal ligation
* Consumes no more than 7 alcoholic beverages per week

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
Change in the area under the curve for urinary estrogen (E1G-AUC) adjusted for cycle length

SECONDARY OUTCOMES:
Effects of exercise on variables known to affect or reflect mitogenic activity as related to breast cancer risk
Changes in other physiologic parameters associated with breast mitotic activity
Extent to which changes in body composition and body mass mediate observed changes in E1G-AUC
Relationship between estrogen and progesterone from daily urinary measurements with observed menstrual cycle alterations (i.e., follicular and luteal phase length changes, and ovulatory status)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Schmitz, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Boyer AL, Arikawa AY, Schmitz KH, Sturgeon KM. Association of Inflammatory Diets with Inflammatory Biomarkers in Women at High Genetic Risk for Breast Cancer. Nutr Cancer. 2022;74(3):816-819. doi: 10.1080/01635581.2021.1986554. Epub 2021 Oct 6. PMID 34615429